CLINICAL TRIAL: NCT04474483
Title: A Pilot Placebo-controlled Randomized Double-blind Trial of Melatonin in Outpatients With COVID-19 Infection
Brief Title: Safety and Efficacy of Melatonin in Outpatients Infected With COVID-19
Acronym: COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficult recruitment and complete first visit in person during thne hight of tne pandemic and later not enough subjects
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Margarita L. Dubocovich, PhD, SUNY Distinguished Professor Dept of Pharmacology and Toxicology, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UBMELCOVID19
Record Dates: First submitted 2020-05-15; First posted 2020-07-16 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: COVID-19
Keywords: Melatonin; COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Melatonin; Methylcellulose; Capsules

STUDY DESIGN:
Intervention Model Description: placebo-controlled randomized double-blind pilot trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Placebo capsules will be prepared with opaque gelatin capsules, filled using methylcellulose and over-encapsulated to appear identical to interventional drug. Placebo capsules will be given orally in the same regimen as intervention (three times daily for 14 days). Capsules will be prepared by the research pharmacist and will be mailed to study subjects directly by courier. Placebo capsules will be stored at room temperature.
  Interventions: Other: Placebo (Methylcellulose) capsule
- Melatonin (Experimental): Melatonin will be administered orally as a 10 mg dose three times a day for 14 days. Size 4 clear vegetable cellulose capsules containing 10 mg melatonin, microcrystalline cellulose, and rice concentrate prepared by Life Extension® will be over-encapsulated in opaque gelatin capsules. Over-encapsulation of melatonin treatments will be done by the research pharmacist and will be mailed to study subjects directly by courier. Melatonin capsules will be stored at room temperature.
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Melatonin will be administered orally as a 10 mg dose three times a day for 14 days. Size 4 clear vegetable cellulose capsules containing 10 mg melatonin, microcrystalline cellulose, and rice concentrate prepared by Life Extension® will be over-encapsulated in opaque gelatin capsules. Over-encapsulation of melatonin treatments will be done by the research pharmacist and will be mailed to study subjects directly by courier. Melatonin capsules will be stored at room temperature.
  Other Names: 5-methoxy-N-acetyl tryptamine
  Arms: Melatonin
Other: Placebo (Methylcellulose) capsule — Placebo capsules will be prepared with opaque gelatin capsules, filled using methylcellulose and over-encapsulated to appear identical to interventional drug. Placebo capsules will be given orally in the same regimen as intervention (three times daily for 14 days). Capsules will be prepared by the research pharmacist and will be mailed to study subjects directly by courier. Placebo capsules will be stored at room temperature.
  Other Names: Methylcellulose
  Arms: Control

SUMMARY:
This study is a pilot randomized, double-blind, placebo-controlled clinical trial to evaluate the safety and efficacy of melatonin in adult outpatients suspected to be afflicted with COVID-19.

DETAILED DESCRIPTION:
This study is a pilot randomized, double-blind, placebo-controlled clinical trial to evaluate the safety and efficacy of melatonin in outpatient adult patients suspected to be afflicted with COVID-19. Participants will be enrolled as outpatients within 72 hrs of onset of COVID-19 symptoms. The study will evaluate the safety of the intervention through 28 days of follow-up as compared to the control arm as assessed by cumulative incidence of serious adverse events (SAEs), cumulative incidence of Grade 3 and 4 adverse events (AEs), and/or discontinuation or temporary suspension of the investigational medication (for any reason). Additionally, the study will aim to evaluate the clinical efficacy of melatonin as compared to placebo as assessed by hospitalization, COVID-19 related symptoms and mortality. The ultimate goal is to determine in an adequately powered study if the anti-inflammatory and antioxidant actions of Melatonin can reduce the severity and prevent progression of COVID-19 when started in mild disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female adult ≥18 years of age at time of enrollment.
* Women of childbearing potential must agree to use at least one primary form of contraception for the duration of the study.
* Subject provides written informed consent prior to initiation of any study procedures.
* Understands and agrees to comply with planned study procedures.
* Agrees to the collection and storage of saliva samples per protocol.

Exclusion Criteria:

* Severe chronic liver disease
* Severe chronic kidney disease or requiring dialysis
* Pregnancy or breast feeding.
* Allergy to the study medication
* Currently taking melatonin
* Currently taking high dose (>500 mg/day) Vitamin C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margarita L Dubocovich, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Background] Aliasgharzadeh A, Farhood B, Amini P, Saffar H, Motevaseli E, Rezapoor S, Nouruzi F, Shabeeb DH, Eleojo Musa A, Mohseni M, Moradi H, Najafi M. Melatonin Attenuates Upregulation of Duox1 and Duox2 and Protects against Lung Injury following Chest Irradiation in Rats. Cell J. 2019 Oct;21(3):236-242. doi: 10.22074/cellj.2019.6207. Epub 2019 Jun 15. PMID 31210428
- [Background] Andersen LP, Gogenur I, Rosenberg J, Reiter RJ. The Safety of Melatonin in Humans. Clin Drug Investig. 2016 Mar;36(3):169-75. doi: 10.1007/s40261-015-0368-5. PMID 26692007
- [Background] Bazyar H, Gholinezhad H, Moradi L, Salehi P, Abadi F, Ravanbakhsh M, Zare Javid A. The effects of melatonin supplementation in adjunct with non-surgical periodontal therapy on periodontal status, serum melatonin and inflammatory markers in type 2 diabetes mellitus patients with chronic periodontitis: a double-blind, placebo-controlled trial. Inflammopharmacology. 2019 Feb;27(1):67-76. doi: 10.1007/s10787-018-0539-0. Epub 2018 Oct 16. PMID 30328031
- [Background] Chen CF, Wang D, Reiter RJ, Yeh DY. Oral melatonin attenuates lung inflammation and airway hyperreactivity induced by inhalation of aerosolized pancreatic fluid in rats. J Pineal Res. 2011 Jan;50(1):46-53. doi: 10.1111/j.1600-079X.2010.00808.x. Epub 2010 Oct 22. PMID 20964706
- [Background] Cheung CY, Poon LL, Ng IH, Luk W, Sia SF, Wu MH, Chan KH, Yuen KY, Gordon S, Guan Y, Peiris JS. Cytokine responses in severe acute respiratory syndrome coronavirus-infected macrophages in vitro: possible relevance to pathogenesis. J Virol. 2005 Jun;79(12):7819-26. doi: 10.1128/JVI.79.12.7819-7826.2005. PMID 15919935
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Kim JY, Lee YD, Kim BJ, Kim SP, Kim DH, Jo KJ, Lee SK, Lee KH, Baik HW. Melatonin improves inflammatory cytokine profiles in lung inflammation associated with sleep deprivation. Mol Med Rep. 2012 May;5(5):1281-4. doi: 10.3892/mmr.2012.814. Epub 2012 Feb 29. PMID 22377793
- [Background] Law HK, Cheung CY, Ng HY, Sia SF, Chan YO, Luk W, Nicholls JM, Peiris JS, Lau YL. Chemokine up-regulation in SARS-coronavirus-infected, monocyte-derived human dendritic cells. Blood. 2005 Oct 1;106(7):2366-74. doi: 10.1182/blood-2004-10-4166. Epub 2005 Apr 28. PMID 15860669
- [Background] Pedreira PR, Garcia-Prieto E, Parra D, Astudillo A, Diaz E, Taboada F, Albaiceta GM. Effects of melatonin in an experimental model of ventilator-induced lung injury. Am J Physiol Lung Cell Mol Physiol. 2008 Nov;295(5):L820-7. doi: 10.1152/ajplung.90211.2008. Epub 2008 Sep 19. PMID 18805959
- [Background] Peng Z, Zhang W, Qiao J, He B. Melatonin attenuates airway inflammation via SIRT1 dependent inhibition of NLRP3 inflammasome and IL-1beta in rats with COPD. Int Immunopharmacol. 2018 Sep;62:23-28. doi: 10.1016/j.intimp.2018.06.033. Epub 2018 Jun 30. PMID 29990691
- [Background] Sanchez-Lopez AL, Ortiz GG, Pacheco-Moises FP, Mireles-Ramirez MA, Bitzer-Quintero OK, Delgado-Lara DLC, Ramirez-Jirano LJ, Velazquez-Brizuela IE. Efficacy of Melatonin on Serum Pro-inflammatory Cytokines and Oxidative Stress Markers in Relapsing Remitting Multiple Sclerosis. Arch Med Res. 2018 Aug;49(6):391-398. doi: 10.1016/j.arcmed.2018.12.004. Epub 2018 Dec 27. PMID 30595364
- [Background] Shang Y, Xu SP, Wu Y, Jiang YX, Wu ZY, Yuan SY, Yao SL. Melatonin reduces acute lung injury in endotoxemic rats. Chin Med J (Engl). 2009 Jun 20;122(12):1388-93. PMID 19567158
- [Background] Shin IS, Park JW, Shin NR, Jeon CM, Kwon OK, Kim JS, Kim JC, Oh SR, Ahn KS. Melatonin reduces airway inflammation in ovalbumin-induced asthma. Immunobiology. 2014 Dec;219(12):901-8. doi: 10.1016/j.imbio.2014.08.004. Epub 2014 Aug 10. PMID 25161126
- [Background] Wang S, Zhao Z, Feng X, Cheng Z, Xiong Z, Wang T, Lin J, Zhang M, Hu J, Fan Y, Reiter RJ, Wang H, Sun D. Melatonin activates Parkin translocation and rescues the impaired mitophagy activity of diabetic cardiomyopathy through Mst1 inhibition. J Cell Mol Med. 2018 Oct;22(10):5132-5144. doi: 10.1111/jcmm.13802. Epub 2018 Jul 31. PMID 30063115
- [Background] Wu GC, Peng CK, Liao WI, Pao HP, Huang KL, Chu SJ. Melatonin receptor agonist protects against acute lung injury induced by ventilator through up-regulation of IL-10 production. Respir Res. 2020 Mar 6;21(1):65. doi: 10.1186/s12931-020-1325-2. PMID 32143642
- [Background] Wu WS, Chou MT, Chao CM, Chang CK, Lin MT, Chang CP. Melatonin reduces acute lung inflammation, edema, and hemorrhage in heatstroke rats. Acta Pharmacol Sin. 2012 Jun;33(6):775-82. doi: 10.1038/aps.2012.29. Epub 2012 May 21. PMID 22609835
- [Background] Zhao X, Sun J, Su W, Shan H, Zhang B, Wang Y, Shabanova A, Shan H, Liang H. Melatonin Protects against Lung Fibrosis by Regulating the Hippo/YAP Pathway. Int J Mol Sci. 2018 Apr 9;19(4):1118. doi: 10.3390/ijms19041118. PMID 29642520
- [Background] Zhang R, Wang X, Ni L, Di X, Ma B, Niu S, Liu C, Reiter RJ. COVID-19: Melatonin as a potential adjuvant treatment. Life Sci. 2020 Jun 1;250:117583. doi: 10.1016/j.lfs.2020.117583. Epub 2020 Mar 23. PMID 32217117

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Melatonin
Started | 3 | 5
Completed | 1 | 3
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Melatonin | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (15.1) | 36.8 (17.4) | 40.8 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Emergent Adverse Events
Description: Evaluate the number of serious adverse effects and discontinuation secondary to toxicity through 28 days of follow-up as compared to the control arm as assessed by: Cumulative number of serious adverse events (SAEs), Cumulative number of Grade 3 and 4 adverse events (AEs), Discontinuation or temporary suspension of the investigational medication (for any reason).
Time Frame: 28 days
Population: All participants who enrolled and took at least one dose of the medication/placebo
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Melatonin
Number analyzed (Participants) | 3 | 5
Participants | 0 | 0

2. Secondary Outcome: Hospitalization
Description: Number of COVID-19 related hospitalizations at 28 days
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Melatonin
Number analyzed (Participants) | 3 | 5
Participants | 1 | 1

3. Secondary Outcome: COVID-19 Related Symptoms
Description: COVID-19 related symptoms (Fever, chills, cough, nasal symptoms, body aches/muscle aches, headache, loss of smell, loss of taste, nausea, vomiting, diarrhea, fatigue, dizziness) that are self-reported and on interview.
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Control | Melatonin
Number analyzed (Participants) | 3 | 5
participants | 3 | 5

4. Secondary Outcome: Rate of Resolution of COVID-19 Related Symptoms
Description: We designed a COVID-19 symptom scale. Participants rated 11 COVID related symptoms on a scale of 0-5. A maximum score of 55 would indicate the worst symptoms, while a score of 0 would indicate no symptoms. Change from baseline (day 1) in the total symptoms score was assessed on days 3, 7, 14, and 28.
Time Frame: 28 days
Population: 1 participant in each group was hospitalized and 1 was lost to follow up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | Melatonin
Number analyzed (Participants) | 3 | 5
score on a scale
  baseline | 23.7 (6.1) | 16.4 (7.7)
  Visit 2: number analyzed (Participants) | 2 | 3
  Visit 2 | 12 (0) | 13.7 (4.2)
  Visit 3: number analyzed (Participants) | 1 | 3
  Visit 3 | 10 | 7.7 (3.5)
  Visit 4: number analyzed (Participants) | 1 | 2
  Visit 4 | 8 | 7.7 (7.1)
  Visit 5: number analyzed (Participants) | 1 | 1
  Visit 5 | 5 | 2

5. Secondary Outcome: Mortality
Description: 28-day mortality
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Melatonin
Number analyzed (Participants) | 3 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Day 1 of enrollment to 6 weeks (42 days) after enrollment.
Description: Information collected at each visit. In 2 participants who were hospitalized, information obtained from family. 2 participants were lost to follow up in spite of repeated attempts to contact them
Arm/Group | Control | Melatonin
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=3) | Melatonin (N=5)
hospitalization (Infections and infestations) | 1 (1) | 1 (1) — COVID-19 progressed leading to hospitalization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT04474483/Prot_SAP_000.pdf